CLINICAL TRIAL: NCT03621657
Title: A Phase II Randomized, Double-blind Placebo-controlled Trial to Determine if Fecal Microbiota Transplantation is Efficacious for Hospitalized Patients With C. Difficile Infection History During Antibiotic Treatment
Brief Title: The GRAFT Study: Gut RecolonizAtion by Fecal Transplantation
Acronym: GRAFT
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Agency for Healthcare Research and Quality (AHRQ) (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2017-0789; A534265 (Other: UW, Madison); SMPH/MEDICINE/INFECT DIS (Other: UW, Madison); 1R03HS025257-01 (AHRQ)
Record Dates: First submitted 2018-07-25; First posted 2018-08-08 (Actual); Results first posted 2021-03-15 (Actual); Last update posted 2021-03-15 (Actual); Status verified 2021-02

CONDITIONS: Clostridium Difficile Infection; C.Difficile Diarrhea; CDI
Keywords: FMT; Fecal Microbiota Transplant
MeSH Terms: conditions — Clostridium Infections | interventions — Fecal Microbiota Transplantation

STUDY DESIGN:
Intervention Model Description: This is a phase 2, double-blind, randomized, placebo-controlled trial assessing the effects of either daily (group 1) or one-time (group 2) oral FMT on the composition and function of gut microbiome compared to placebo (group 3) in a population of patients with a history of Clostridium difficile infection (CDI).
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Low dose FMT Capsule DE (Experimental): FMT Capsule double-encapsulated (DE) by mouth, 5 capsules once daily with antibiotic, followed by 5 capsules daily for 7 days post-antibiotic
  Interventions: Drug: Low Dose FMT Capsule DE
- Single dose FMT Capsule DE (Active Comparator): FMT Capsule DE by mouth, 30 capsules in a single one-time dose 48-72 post-antibiotic course.
  Interventions: Drug: Single Dose FMT Capsule DE
- Placebo Oral Capsule (Placebo Comparator): Oral placebo capsules manufactured to mimic study capsule, 5 capsules daily with antibiotic course, followed by 5 capsules for 7 days post-antibiotic
  Interventions: Drug: Placebo oral capsule

INTERVENTIONS:
Drug: Low Dose FMT Capsule DE — 5 FMT Capsule DE along with antibiotic; followed by five capsules FMT Capsule DE x 7 days post-antibiotic course.
  Other Names: FMT Capsule DE
  Arms: Low dose FMT Capsule DE
Drug: Single Dose FMT Capsule DE — 30 pill FMT Capsule DE treatment x 1, 48-72 hours following completion of antibiotic treatment.
  Other Names: FMT Capsule DE
  Arms: Single dose FMT Capsule DE
Drug: Placebo oral capsule — Five capsules per day along with antibiotic; followed by five capsules per day for seven days post-antibiotic treatment.
  Other Names: Placebo
  Arms: Placebo Oral Capsule

SUMMARY:
The primary objective of this study is to compare the gut microbiota and clinical outcomes of oral FMT during antibiotic treatment, immediately following antibiotic treatment, and placebo. The second objective is to assess the safety and feasibility of daily oral Fecal Microbiome Transplant (FMT) as a treatment option.

DETAILED DESCRIPTION:
Clostridium difficile is the most frequent bacterial cause of antibiotic-associated diarrhea. Those with a previous C. difficile infection (CDI) are at high risk of recurrent infection. Recurrent CDI often occurs when the normal gut microbiota are disrupted. Dysbiosis of the gut microbiota predisposes to CDI which, despite treatment can recur in 30% of patients. A novel way to prevent CDI recurrence is by instilling feces from a healthy individual into the intestine of the CDI patient, thereby restoring balance in the gut microbiota. However, it is unknown whether or not fecal microbiota transplantation (FMT) is an efficacious choice for CDI recurrence prevention when used concurrently with antibiotics. We propose a pilot randomized, double-blind placebo controlled trial comparing oral FMT with placebo in patients with a history of CDI, currently undergoing antibiotic treatment. We will collect fecal samples from subjects prior to, during, and after FMT and collect metagenomics and microbiologic data on microbiota composition and function, and CDI recurrence. The trial's primary outcome is gut microbial composition and function. Secondary outcomes are feasibility and safety, and recurrent CDI during the trial period. In this 3 group study, FMT will be administered daily via oral capsules containing frozen fecal microbiota from universal donors in group 1, administered at the end of antibiotic treatment for group 2, and group 3 will receive daily placebo. The results of this study will provide the necessary pilot data to examine whether or not concurrent FMT in antibiotic treated patients who are at high risk for recurrent CDI can maintain a diverse healthy GI microbiota.

ELIGIBILITY:
Inclusion Criteria:

1. Cognitively intact and willing to provide informed consent
2. Willing and able to comply with all study procedures for the duration of the study
3. Able to take oral medications
4. Age 18 or over
5. Recent CDI episode occurring in the last 180 days with completion of therapy as confirmed by the electronic medical record (EMR)
6. Receiving antibiotics at enrollment for reasons other than CDI and having taken the antibiotics for no longer than 10 days.
7. Women of childbearing potential in a sexual relationship with men must use an acceptable method of contraception (including, but not limited to, barriers with additional spermicidal foam or jelly, intrauterine devices, hormonal contraception started at least 30 days before enrollment into the study, or intercourse with men who underwent a vasectomy) for 4 weeks following completion of the study treatment,
8. Males must agree to avoid impregnation of women during and for 4 weeks following completion of the study treatment.
9. Able to take the test capsule successfully with no signs or symptoms of dysphagia.

Exclusion Criteria:

1. Females who are pregnant, lactating, or planning to become pregnant during the study. Female patients of childbearing potential will take a pregnancy test at the intervention visit and will be excluded if pregnant.
2. Inability (e.g. dysphagia) to or unwilling to swallow capsules
3. Known or suspected toxic megacolon and or known small bowel ileus
4. Bowel obstruction or other gut motility issues occurring in the last two weeks taht are unresolved as noted by the patient or in the EMR
5. Major gastrointestinal surgery (e.g. significant bowel resection) within 3 months before enrollment not including appendectomy or cholecystectomy.
6. History of bariatric or colectomy surgery
7. Concurrent intensive induction chemotherapy, radiation therapy, or biologic treatment for an active malignancy. Patients on maintenance chemotherapy may be enrolled after consultation with the medical monitor.
8. Expected life expectancy less than 6 months.
9. Patients with severe anaphylactic or anaphylactoid food allergy.
10. Solid organ transplant recipients ≤90 days post-transplant or on active treatment for rejection
11. Neutropenia (≤500 neutrophils/mL) or other severe immunosuppression. Anti-tumor necrosis factor (TNF) will be permitted. Patients on monoclonal antibodies to B and T cells, glucocorticoids, antimetabolites (azathioprine, 6-mercaptopurine, methotrexate), calcineurin inhibitors (tacrolimus, cyclosporine), and mycophenolate mofetil may only be enrolled after consultation with the medical monitor.
12. At risk of CMV/EBV associated disease, negative immunoglobulin gamma (IgG) testing for cytomegalovirus (CMV) or Epstein Barr Virus (EBV)
13. Any other gastrointestinal illness including diarrhea
14. On oral vancomycin or metronidazole
15. Having been taking the currently prescribed antibiotic for over 10 days
16. Any condition that would jeopardize the safety or rights of the patient, would make it unlikely for the patient to complete the study, or would confound the results of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2020-02-27 (Actual); Study Completion 2020-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nasia Safdar, MD, PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital & Clinics, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Low Dose FMT Capsule DE | Placebo Oral Capsule | Single Dose FMT Capsule DE
Started | 0 | 0 | 1
Completed | 0 | 0 | 1
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Study was completed with only 1 participant enrolled.
Groups:
- Total: Total of all reporting groups
Arm/Group | Low Dose FMT Capsule DE | Placebo Oral Capsule | Single Dose FMT Capsule DE | Total
Number analyzed (Participants) | 0 | 0 | 1 | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 0 | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 0 | 0 | 1 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 0
  Not Hispanic or Latino | 0 | 0 | 1 | 1
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 0 | 0 | 1 | 1
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Assess Efficacy of Oral FMT on Composition and Function of the Gut Microbiota Compared to Placebo.
Description: Assess microbial composition of stool using 16s targeted sequencing and shotgun metagenomics
Time Frame: 60 days
Population: There are no results due to low enrollment (N=1).
Arm/Group | Low Dose FMT Capsule DE | Placebo Oral Capsule | Single Dose FMT Capsule DE
Number analyzed (Participants) | 0 | 0 | 0

2. Secondary Outcome: Comparison of Treatment-related Adverse Events in the Oral FMT Regimens Versus Placebo.
Description: Proportion of participants with treatment-related adverse events as assessed by CTCAE v4.0, including serious adverse events, will be assessed. We will also assess proportion of newly diagnosed infectious diseases, which are considered adverse events of special interest (AESI) after randomization.
Time Frame: 60 days
Population: There are no results due to low enrollment (N=1)
Arm/Group | Low Dose FMT Capsule DE | Single Dose FMT Capsule DE | Placebo Oral Capsule
Number analyzed (Participants) | 0 | 0 | 0

3. Secondary Outcome: Determine the Rate of Clostridium Difficile Infection (CDI) During Oral FMT Regimens Versus Placebo
Description: Collection of CDI infection rates from baseline to end of study and comparison between both oral FMT groups versus placebo.
Time Frame: 60 days
Population: There are no results due to low enrollment (N=1)
Arm/Group | Low Dose FMT Capsule DE | Single Dose FMT Capsule DE | Placebo Oral Capsule
Number analyzed (Participants) | 0 | 0 | 0

4. Secondary Outcome: Evaluate Time to Clostridium Difficile Infection (CDI) and/or Colonization With C. Difficile.
Description: C. difficile colonization will be detected in stool samples submitted at baseline through end of study. If patients' become colonized, time from randomization to colonization is collected. Comparisons are made between the oral FMT groups and placebo.
Time Frame: 60 days
Population: There are no results due to low enrollment (N=1)
Arm/Group | Low Dose FMT Capsule DE | Single Dose FMT Capsule DE | Placebo Oral Capsule
Number analyzed (Participants) | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: 6 months
Description: Insufficient participant population, low enrollment
Arm/Group | Low Dose FMT Capsule DE | Placebo Oral Capsule | Single Dose FMT Capsule DE
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/1
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 1/1
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Low Dose FMT Capsule DE (N=0) | Placebo Oral Capsule (N=0) | Single Dose FMT Capsule DE (N=1)
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) — Basal cell carcinoma, unrelated to study procedures, resolved without sequelae

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-12-05): https://cdn.clinicaltrials.gov/large-docs/57/NCT03621657/Prot_SAP_000.pdf